CLINICAL TRIAL: NCT05336292
Title: Acceptability and Preliminary Results of a Meaning-focused Intervention in the Army: A Case Series Study. Assessment of Meaningful Life Intervention in the Spanish Forces
Brief Title: Meaning-focused Intervention in the Army
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UComplutenseMadrid-Meaningful
Record Dates: First submitted 2022-03-17; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Meaningful Life
Keywords: Meaningful life; Meaningful at work; Propose; Well-being; Emotional regulation
MeSH Terms: conditions — Emotional Regulation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups; intervention based on meaningful life(MLI); intervention based on meaningful life and emotional regulation (MLI+ER) or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meaningful life intervention (Active Comparator): We will work with psychological skills, meaningful life model, mindfulness skills ,personal values, the Wellbeing Model (Ryff, 1989) . The strengths of character (Park et al., 2004) and sources meaningful life. We will identify ways to use strengths and enhance meaningful life and develop an action plan to improve strengths. ). To identify the Meaning at the work. Link our strengths and values to our goals and purposes. Apply the SMART Method to achieve meaningful goals. Visualizing Our Best Future Self (Burton & King, 2004).
  Interventions: Behavioral: Meaningful life-focused intervention; Behavioral: Meaningful life and emotional regulation-focused intervention; Behavioral: Control Group
- Meaningful life and emotional regulation (Active Comparator): Program Based on meaningful life and Emotional Regulation (MLI+ER) Session 1 Emotional regulation as a path towards the meaningful life Mindfulness training (emotional mindfulness) Generate knowledge of emotions and their functioning Session 2 Emotional Psychoeducation Emotional care To Know the well-being model Carol Ryff and Vital Sense To Understand the process of emotional regulation Session 3 Strengths and Personal Values Cultivate introspection and self-knowledge (Mindfulness, Carlson, 2013; Klussman, 2020) To Know the strengths of character (Park et al., 2004) and sources of vital meaning Identify ways to use strengths and enhance the sense of life Making Core Values Real (My 80th Birthday Speech; Harris, 2009) Note: Sessions 4, 5 and 6 are the same as the intervention based on meaningful life
  Interventions: Behavioral: Meaningful life-focused intervention; Behavioral: Meaningful life and emotional regulation-focused intervention; Behavioral: Control Group
- Control group (Active Comparator): The waiting list will be the control group. Participants will not be part of the program. They will participate in a day of positive psychology
  Interventions: Behavioral: Meaningful life-focused intervention; Behavioral: Meaningful life and emotional regulation-focused intervention; Behavioral: Control Group

INTERVENTIONS:
Behavioral: Meaningful life-focused intervention — The intervention works different skills to increase the meaningful life in the general population and specifically in the army.
Behavioral: Meaningful life and emotional regulation-focused intervention — The intervention works different skills to increase the meaningful life and emotional regulation in the general population and specifically in the army.
Behavioral: Control Group — This group does not do any intervention

SUMMARY:
The purpose of this research is to contribute to the empirical study of meaningful life interventions in the general population, since it is a sample of active professionals. To get the research objectives, two studies are proposed.

In the present investigation the effects of two interventions in meaningful life will be analyzed and will be compared with a control group. The first group will be an intervention based on meaningful life (MLI), the second group an intervention based on meaningful life and emotional regulation (MIL+ER) and the third group will be a control group on the waiting list. The assignment will be random and both programs will consist of six sessions, once a week, of 120 minutes.

Prior to the main study, a pilot study will be carried out with the aim of describing the possible individual benefits of the meaningful life intervention, and at the same time analyzing whether emotional regulation favors meaningful life. The acceptability and feasibility of both programs will also be evaluated.

DETAILED DESCRIPTION:
The structure of the program will include tools for the promotion of meaning through the understanding of oneself, the practice of mindfulness, strengths, values, analysis of objectives and action plans to achieve them . In the MLI+ER group, training in emotional regulation skills will be included as an element that enhances the meaning of life, as suggested by some studies.

Objectives and hypotheses Studio 1

The investigators set ourselves the following objectives:

1. Explore the feasibility of enhancing the sense of life and work through an intervention based on the sense of life.
2. To explore the usefulness of an emotional regulation component in an intervention based on a meaningful life to enhance the effects on a meaningful life and a meaningful at work.
3. To explore the possible impact of an intervention based on meaningful life in other relevant aspects such as meaningful at work, burnout, work commitment, well-being, emotional dysregulation and depression
4. Check if an intervention based on meaningful life is acceptable and feasible in a non-clinical population in the military context.
5. Explore aspects to improve in the protocol based on the quantitative and qualitative results.

Study 2 Objectives: To compare the effects of a MLI-based intervention compared to a combined MLI+ER program and to analyze its impact on subjective well-being, emotional regulation, depressive symptomatology, burnout, and work commitment, as well as the mechanisms of change.

Hypothesis 1: The intervention group MLI and ER+MLI will present higher scores in meaningful life and meaningful at work after the intervention with respect to the subjects of the control group.

Hypothesis 2: The MLI and MLI+ER intervention group will present higher scores in subjective well-being, emotional regulation, depressive symptomatology, burnout and work commitment (secondary indicators) after the intervention compared to the control group subjects.

Hypothesis 3: Compared to the MLI group, the MLI+ER group will show greater increases in well-being (i.e., PHI subscale), emotional regulation, and meaningful life after the intervention.

Hypothesis 4: Participants in both interventions will show high levels of acceptability and satisfaction with the intervention.

The sample of this research will be workers of the Spanish Armed Forces, once the project is approved by the Research Ethics Committee of the Complutense University of Madrid. Participants will sign an informed consent form and receive an information sheet with the purpose of the research before starting the intervention.

The pilot study will be carried out with the first 18 participants in the program, being excluded from the total expected sample size. The estimated sample size is made from the G-Power 3.1 software, taking as a reference the effect size of 0.37 suggested by the literature on the effect of Mindfulness interventions on the vital sense (Chu, 2020). The investigators take a conservative approach, adopting an effect size of 0.30 which may correspond according to Cohen (d) to a medium-moderate effect size. The expected total sample size will be 120 participants.

The participants will be recruited voluntarily in a Military Unit in Madrid. Talks will be held between potential participating staff. Volunteers will register through their offices, in turn, the registration will be sent by organic chain to our department. Once the request of the interested personnel has been made, participants will be contacted via email or telephone. Participants will fill in all the pre, post and follow-up measures (via google forms) and will be randomly assigned to one of the three groups; intervention based on meaningful life (MLI); intervention based on meaningful life and emotional regulation (MLI+ER) or control group. Once assigned to the group, the program will begin with six sessions, once a week, for 120 minutes.

The design proposed to achieve the first objective will be a qualitative case study in order to investigate the individual effects at two moments: pre-post intervention, in the set of measures described above and in the five questions to evaluate individual satisfaction with the program. It will be carried out with the first 18 participants who complete the program and will form part of the pilot study.

For the rest of the objectives included in the second study, the proposed design is experimental with random assignment to the three groups; the two intervention modalities and control group. Repeated measures will be applied in three moments, pre and post and follow-up at 4 months. At the end of the data collection of all the participants, there will be a sample of 120 participants (excluding the 18 participants of the pilot study); (MLI) n= (40), (MLI+ER) n= (40) and (CG) n= (40). A quantitative and qualitative research design will be adopted to investigate the satisfaction, acceptability and feasibility of the program through the post measures and degree of acceptability-satisfaction with the intervention (CSQ-8).

Given the conditions of the size of the sample and to control the variability due to other factors, such as the programming of activities in the organization. The personnel will be organized randomly, in groups of 8 people in each modality, distributed in seven shifts of six sessions. In each turn, the two modalities will be carried out at the same time, in addition to their control group. This is justified by the type of sample and the conditions of the organization.

Regarding the analysis techniques provided for in the first study, a descriptive analysis of the mean of the first participants will be carried out, in addition to the non-parametric tests and qualitative analysis of the satisfaction comments. For the second study, once the data collection is finished, the pertinent tests of homoscedasticity and normality tests will be carried out to check if the data are parametric, and thus be able to use parametric techniques. In this case, the tests used would be: normality tests, group equivalence, Anova for repeated measures, Anova for independent samples, Regression analysis to evaluate the predictive capacity of the variables.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the research will be active military personnel, or an active worker, over 18 years of age.

Exclusion Criteria:

* The exclusion criteria will be being on medical or psychiatric leave or having a significant level of depression (PHQ greater than or equal to 10). People excluded for this reason will be referred to a psychological care service.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-13 (Estimated)

PRIMARY OUTCOMES:
Change in Meaningful life | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Meaningful life Questionnaire; MLQ de Steger M., 2006, It is a 10-item instrument with two subscales that measure presence and the search for meaning in life. Items are rated on a Likert scale from 1 (Absolutely false) to 7 (Absolutely true). A minimum score of 24 points on each subscale reflects higher levels of presence and search for meaning in life, respectively.
Change in Meaningful at work | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Work and Meaningful Inventory; WAMI, Steger M., 2012; It is a 10-item instrument. It measures the perception that the individual has about the meaning of his work. The WAMI contains 3 subscales: positive meaning at work (PM), feeling that the work one does is important, creating meaning through work (MM), building meaning in one's personal life through what one does at work job; and great motivations towards others (GG), believing that work benefits and does good for others and society in general. Each item is evaluated on a Likert-type scale ranging from 1 (Absolutely false) to 5 (Absolutely true). The total score ranges from 10 to 50, the higher the score, the more meaning experienced through the work.
Change in Well-being | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Pemberton happiness index; Vazquez C. y Hervas G., 2013; This scale is a measure of well-being that integrates hedonic and eudaimonic aspects. The scale contains 11 items of remembered well-being and 10 items of experienced well-being. The sum of these scales results in a well-being index. The recalled well-being scale has a Likert scale ranging from 0 (completely disagree) to 10 (completely agree). The well-being index has a score from 0 to 10.

SECONDARY OUTCOMES:
Change in Burnout | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Maslach Burnout Inventory (MBI; Maslach & Jackson, 1981; Spanish version Bresó, et al., 2007). It measures the degree of burnout. It is a 15-item instrument. It is assessed on a Likert-type frequency scale that ranges from 0 (never) to 6 (always). It consists of three scales: five items evaluate exhaustion, four items evaluate cynicism, and six items evaluate professional efficacy.
Change in Engagement at work | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Ultrech Work Engagement Scale (UWES-9; Schaufeli & Bakker, 2003; Spanish adaptation; Schaufeli et al., 2006) includes 9 items that reflect the three dimensions of work engagement. Each item is evaluated on a Likert-type scale ranging from 0 (never/never) to 6 (always/every day). Each scale contains 3 items. The scales are vigor, dedication and absorption, in our study we work with the total scale from 0 to 6.
Change in Emotional regulation | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Difficulties in Emotion Regulation Scale (DERS; de Gratz and Roemer, 2004; Spanish adaptation of Hervás & Jódar, R., 2008). This scale evaluates the deficit that exists for optimal emotional regulation through 28 items. The responses are 5-point Likert-type (from "Almost never/0-10% of the time" to "Almost always/90-100% of the time). Although the scale has 5 factors: Emotional lack of control (lack of access to effective emotion regulation strategies (strategies) and lack of ability to manage one's impulses during negative emotions (impulse) ; Emotional confusion (lack of clarity about the nature of one's emotions (clarity ), Everyday interference (lack of ability to engage in goal-directed activities during negative emotions (goals), Emotional neglect (lack of awareness of one's emotions (awareness) and Emotional rejection (lack of acceptance of one's emotions (nonacceptance). In this study, the Total Emotional Dysregulation Scale was used with a score of 28 to 140.
Change in Depression after intervention | "pre intervention", "immediately after intervention" and "4 months after the end of the intervention"
  Patient Health Questionnaire (PHQ-9; Kroenke et al, 2001; Diez-Quevedo et al., 2001) is an instrument that contains 9 items. It is based on the diagnostic criteria of the DSM-IV and measures the severity of depression. The 9 articles are scored with a score of 4 points. The score ranges from 0 = "not at all" to 3 = "almost every day". The cut-off points for mild depression are 5, moderately 10, moderately severe 15, and severe 20.
Client Satisfaction Questionnaire after intervention and open questions | "immediately after intervention"
  The score goes from 8 to 32. Range of Dissatisfied or less satisfied (8-16), Satisfied (17-30), Very satisfied (31-32). Open questions : Do you consider that the content you worked on has helped you clarify the things that are important and valuable in your life? Do you consider that the content you worked on has helped you find meaning in what you do at work and improve your well-being at work? Do you think that the content worked on has helped you clarify the things that are important and valuable in your life? , A third element with a Likert-type scale evaluates the effect of the program on personal well-being. In general, do you consider that the program can be useful to improve your personal well-being? Finally, participants are asked four open questions, inviting them to evaluate and make suggestions to improve the program

CONTACTS AND LOCATIONS:
Locations (1):
- Militaries units, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request, due to the provenance of the sample.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the data collection and analysis is finished, they can be facilitated and shared for justified reasons during the time deemed appropriate, due to the characteristics of the sample.
Access Criteria: The data will be available upon reasonable request, due to the provenance of the sample.

REFERENCES:
- [Background] Chu, S., & Mak, W. (2020). How Mindfulness Enhances Meaning in Life: A Meta-Analysis of Correlational Studies and Randomized Controlled Trials. Mindfulness. 11, 177-193 https://doi.org/10.1007/s12671-019-01258-9.
- [Background] Hicks, J., & King, L. (2009). Positive mood and social relatedness as information about meaning in life. The Journal of Positive Psychology, 4(6), 471-482. https://doi.org/10.1080/17439760903271108.
- [Background] Martela, F., & Steger, M. (2016). The three meanings of meaning in life: Distinguishing coherence, purpose and significance. The Journal of Positive Psychology, 11, 531-45.
- [Background] Ryff, C. (1989).
- [Background] Steger, M., Dik, B., & Duffy, R. (2012). Measuring meaningful work: The work and Meaning Inventory (WAMI). Journal of Career Assesment, 20, 322-37.
- [Background] Steger, M., Frazier, P., Oishi, S., & Kaler, M. (2006). The Meaning in Life Questionnaire: Assesing the Presence of and Search for Meaning in Life. Journal of Counselling Psychology, 53, 1, 80-93. DOI: 10.1037/0022-0167.53.1.80.
- [Background] Schaufeli, W. B., Bakker, A. B., & Salanova, M. (2006). The measurement of work engagement with a short questionnaire. A cross-national study. Educational and Psychological Measurement, 66, 701-716. https://doi.org/10.1177/0013164405282471.
- [Background] Park, N., Peterson, C., & Seligman, M. E. (2004). Strengths of character and well-being. Journal of social and Clinical Psychology, 23(5), 603-619. https://doi.org/10.1521/jscp.23.5.603.50748
- [Background] Maslach, C. & Jackson, S.E. (1981), The measurement of experienced burnout. J. Organiz. Behav., 2: 99-113. https://doi.org/10.1002/job.4030020205
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hervás, G., & Jódar, R. (2008). Adaptación al castellano de la Escala de Dificultades en la Regulación Emocional The spanish version of the Difficulties in Emotion Regulation Scale. Clínica y Salud, 19(2), 139. https://psycnet.apa.org/record/2008-17752-001
- [Background] Harris, R. (2009). ACT Made Simple: An easy-toread primer on Acceptance and Commitment Therapy. Oakland: CA: New Har
- [Background] Burton, CM & King, LA. 2004. The health benefits of writing about intensely positive experiences. Journal of Research in Personality, 38: 150-163. https://doi.org/10.1016/S0092-6566(03)00058-8
- [Background] Shin, J., & Steger, M. (2014). Promoting Meaning and Purpose in Life. En A. C. Parks, S.M. Schueller. The Wiley-Blackwell Handbook of Psychology of Positive Psychological Interventions, First Edition. London: Willey-Blackwell.
- [Background] Wong, P. (2010). Meaning therapy: an integrative and positive existential psicotherapy. Journal of Contemporary Psicotherapy, 40, 85-93.
- [Background] Steger, M. (2017). Creating Meaning and Purpose in Work. In L. Oades, M.F. Steger, A. Della Fave, and J. Passmore, (eds.), The Wiley-Blackwell Handbook of Psychology of Positive and Strenghts-based Approacheas at work, pp. 60-81. London: Willey-Blackwell.
- [Background] Miao M, Gan Y. How does meaning in life predict proactive coping? The self-regulatory mechanism on emotion and cognition. J Pers. 2019 Jun;87(3):579-592. doi: 10.1111/jopy.12416. Epub 2018 Aug 5. PMID 29999537
- [Background] Steger, M., & Ekman, E. (2016). Working it: Making meaning with workplace mindfulness. In: Mindfulness and positive psychology. New York: Itzvan; 2016:1-29.
- [Background] Carlson EN. Overcoming the Barriers to Self-Knowledge: Mindfulness as a Path to Seeing Yourself as You Really Are. Perspect Psychol Sci. 2013 Mar;8(2):173-86. doi: 10.1177/1745691612462584. PMID 26172498
- [Background] Park, N., Park, M. &Peterson, C. (2010), When is the Search for Meaning Related to Life Satisfaction? Applied Psychology: Health and Well-Being, 2: 113. https://doi.org/10.1111/j.1758-0854.2009.01024.x
- Available data/document: Individual Participant Data Set — https://drive.google.com/drive/folders/1Z6K71rEcfJHXIzsurwREdgHRweFwgFW3 — Data will be made available upon reasonable request